CLINICAL TRIAL: NCT02827760
Title: The Effect of Prebiotic Synergy1 Supplementation on Microbiota, Protein Metabolism and Gastrointestinal (GI) Symptoms in People Consuming High Protein Diet
Acronym: ITF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Xuedan Wang, PhD candidate, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IFTPRO00
Record Dates: First submitted 2016-06-14; First posted 2016-07-11 (Estimated); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Gut Microbiota
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Maltodextrin DE19 (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Maltodextrin
- Prebiotic Synergy1 (Active Comparator): Effective prebiotic
  Interventions: Dietary Supplement: Synergy1

INTERVENTIONS:
Dietary Supplement: Synergy1 — Inulin type fructans
  Arms: Prebiotic Synergy1
Dietary Supplement: Maltodextrin
  Arms: Maltodextrin DE19

SUMMARY:
The composition and metabolism of human gut microbiota play crucial roles in health. Microbial colonisation of the gastrointestinal tract varies widely, with the large intestine having not only the highest density of microbes in terms of bacterial cells per gram but also the most metabolically active microbial community. Genetics, mode of birth, infant feeding patterns, antibiotic usage, sanitary living conditions and long term dietary habits contribute towards shaping the composition of the gut microbiome. Diet clearly has a major impact on variation in the gut microbiota composition, and this can be detected in faecal samples after only a few days. The bacterial metabolism of dietary components produces much chemical diversity in the large intestine with protective or detrimental effects on disease development.

Dietary protein levels are relatively high in western European populations, up to 103g/d, as reported by Food and Agriculture Organization. This may result in high levels, entering the large gut where it can become a substrate for proteolytic bacteria. Protein specifically can provide nutrition for microorganisms but metabolites from bacterial protein breakdown can be detrimental. Protein intake from the diet might not be the only source of microbial proteolysis; the human body also secretes considerable amounts of protein into the digestive lumen which can potentially be used by the microflora. On the contrary, end products of carbohydrate metabolism can be positive for health. In this context, prebiotics are carbohydrates that are resistant to digestion and can become available for bacteria in the colon to produce short chain fatty acids and inhibit the production of harmful metabolites. A switch towards more carbohydrate metabolism in the colon, at the expense of proteolysis therefore has positive capacity through the production of more benign metabolites.

Rationale for design Prebiotics are dietary ingredients that target carbohydrate digesting bacteria only. Given the high intake levels of protein in Western populations, they may be useful to modulate the composition/activity of the microbial gut ecology for improved health.

Among prebiotic nutrients, inulin-type fructans (ITF) are well characterized and their administration promotes growth of beneficial microorganisms like Bifidobacterium spp. .These microorganisms are involved in the reduction of intestinal endotoxin concentration, improve glucose tolerance, exert benefits upon immune function and inhibit pathogens. In healthy individuals, ITF intake promotes satiety and modulates gut peptides regulating food intake.

The aim of the present study is to investigate the effect of inulin-type fructans (ITF) on the negative consequences of colonic fermentation in individuals consuming high protein diets. The hypothesis to be tested is that their action promotes carbohydrate degrading bacteria at the expense of protein utilisers.

ELIGIBILITY:
Inclusion Criteria:

* In good general health.
* Having high protein diet.
* The volunteer has given written informed consent to participate and is willing to participate in the entire study.

Exclusion Criteria:

* History or evidence of intestinal disease; such as tumour, Irritable Bowel Syndrome, etc., within the previous 5 years.
* Received antibiotics in the previous six months
* Not willing to cease the consumption of probiotic or prebiotic preparations for the duration of the study
* Former participation in another study involving prebiotic or probiotic preparations within the previous 2-weeks, or intention to use such products during the course of the study (please note sensory evaluations may be still permitted after discussion with the Investigator)
* History of malignancy within the previous 5 years (with exception of well-treated basal cell carcinoma or in situ cervical carcinoma).
* Diabetes
* Smoker
* Lactose intolerant
* Allergic to gluten
* Currently prescribed immunosuppressive drugs.
* Participants will be required to withdraw should they begin taking any of the ineligible medication.
* Intention to use regularly other medication which affects gastrointestinal motility.
* History of alcohol or drug misuse.
* Using statins
* Suffer from any major conditions involving the following: Head, Ears, Eyes, Nose and Throat, Dermatological/Connective tissue, Neurological, Lymphatic, Urogenital/Rectal, Abdominal, Respiratory, A previous cardiovascular event within the last 6 months, presence of secondary dyslipemia related to thyroid dysfunction, used any drug affecting lipid metabolism in previous 3 months, a history of alcohol abuse.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Changes on the faecal microbiota composition by fluorescence in situ hybridisation | 12 months
  Changes in faecal bacterial populations will be assessed through the use of fluorescence in situ hybridisation with molecular probes targeting 16S rRNA genes. Genotypic probes targeting the predominant components of the gut microflora (Bacteroides, Bifidobacterium, Clostridium, Lactobacillus, Eubacterium, Atopobacterium, sulphate reducing bacteria and enterobacteria) and total bacteria will be tagged with fluorescent markers such that quantifiable changes may be determined.
Effect on faecal microbiota activity using NMR | 12 months
  Relative abundance of various metabolites will be analysed by Nuclear magnetic resonance spectroscopy (NMR).
Changes in faecal water short chain fatty acids (SCFAs) using gas chromatography | 12 months
  Concentrations of short chain fatty acids (SCFAs) will be quantified using gas chromatography (GC).

SECONDARY OUTCOMES:
Daily assessment of stools consistency | 12 months
  Stool consistency will be scored based on Bristol chart.
Daily assessment of gastrointestinal symptoms | 12 months
  Number of abnormal pain, bloating or flatulence will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Food and Nutritional sciences, Reading, Berkshire, United Kingdom